CLINICAL TRIAL: NCT05222334
Title: Perioperative Respiratory and Analgesic Effects of Ultrasound-Guided Extrafascial Versus Intrafascial Interscalene Brachial Plexus Block in Patients Undergoing Shoulder Arthroscopy
Brief Title: Ultrasound-Guided Extrafascial Versus Intrafascial Interscalene Brachial Plexus Block in Shoulder Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Radwa Emad Eissa, Assistant lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 33802/4/20
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Arthroscopy; Analgesia; Intrafascial Interscalene Brachial Plexus Block
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrafascial interscalene brachial plexus block group (Experimental): The patients will receive 10 ml of 0.5% bupivacaine for intrafascial interscalene brachial plexus block group
  Interventions: Procedure: Intrafascial interscalene brachial plexus block; Drug: Bupivacaine
- Extrafascial interscalene brachial plexus block group (Experimental): The patients will receive 10 ml of 0.5% bupivacaine for extrafascial interscalene brachial plexus block group
  Interventions: Procedure: Extrafascial interscalene brachial plexus block group; Drug: Bupivacaine

INTERVENTIONS:
Procedure: Intrafascial interscalene brachial plexus block — After sterilization of skin with povidone-iodine (betadine) and skin infiltration with 1-3ml lidocaine 1%, interscalene brachial plexus block will be performed using an ultrasound machine (Phillips Cx-50,Amsterdam, Netherlands) with a linear probe (L12-3 MHz) will be used in both groups. The US transducer will be placed under aseptic fashion on the lateral side of the neck at the cricoid cartilage level to view three hypoechoic structures, that represent the roots of the brachial plexus.
  The two outermost nerve roots (C5 and C6) between the anterior and the middle scalene muscles will be identified and the local anesthetic (10 ml 0.5% bupivacaine) is then injected, so that spread will be seen immediately between the C5 and the C6 nerve roots.
  Arms: Intrafascial interscalene brachial plexus block group
Procedure: Extrafascial interscalene brachial plexus block group — Final needle tip position will be 4 mm lateral to the brachial plexus sheath, at a level equidistant between C5 and C6 roots. The distance of 4 mm is chosen according to the calculated success rate over 90% reported. the local anesthetic (10 ml 0.5% bupivacaine) is then injected
  Arms: Extrafascial interscalene brachial plexus block group
Drug: Bupivacaine — bupivacaine

SUMMARY:
The aim of the study is to compare the diaphragmatic excursion and postoperative analgesia in the extrafascial versus intrafascial Interscalene brachial plexus block in patients undergoing shoulder arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both sexes aged (21-60years) with American Society of Anesthesiologists (ASA) physical status I/II scheduled for shoulder arthroscopy

Exclusion Criteria:

1. Patient refusal.
2. Pre-existing (obstructive or restrictive) pulmonary disease.
3. Bleeding disorders (coagulopathy).
4. Mental dysfunction.
5. History of allergy to local anesthetics.
6. Pregnancy
7. Body mass index (BMI) >40

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of diaphragmatic excursion reduction after interscalene block | 30 min postoperative.
  The diaphragmatic excursion will be measured before the procedure (pre-block), 30 min after the block, and postoperative in Post-Anesthesia Care Unit. Hemidiaphragmatic paresis is defined as hemi-diaphragmatic excursion reduction superior to 75% compared with the pre-procedure value.

SECONDARY OUTCOMES:
Efficacy of block (sensory) | 30 minutes Postoperatively
  The sensory block is assessed by pinprick on a score ranging from 2 to 0 scored as full sensation =2, decreased sensation =1, and loss of sensation to touch or pinprick=0. A successful block is defined as complete sensory (score= 0) in the distribution of the C5 and C6 nerve roots within 30 min of performing the Interscalene Brachial Plexus Block.
Forced expiratory volume in 1 second (FEV 1) | Intraoperatively or 30 minutes postoperatively
  Respiratory related outcome: pulmonary function test including forced expiratory volume in 1 second (FEV 1) will be assessed before block and 30 minutes after discharge to Post-Anesthesia Care Unit (PACU) with a laboratory spirometer (Carevusion Germany Spirometer; Master screen PFT). The best value will be measured and recorded
Pain score using numerical rating scale (NRS) | 24 hours Postoperative
  Numerical rating scale (NRS) for assessment of pain intensity (0 = no pain) to (10 = intolerable pain), pain relief is defined as a numerical rating scale of 3 or lower. If the score is >3, the patient will need analgesia in the form of morphine 0.05 mg/kg till it decreases to ≤3. numerical rating scale will be assessed and recorded on arrival to Post-Anesthesia Care Unit (PACU), 1, 2, 4, 8, 12, and 24 hr postoperatively by an anesthesiologist who is blinded to the study groups
Total postoperative analgesic consumption | 24 hours Postoperative
  Total consumption of rescue analgesia in form of morphine 0.05 mg/kg/ dose will be recorded
Peak expiratory flow (PEF) | Intraoperatively or 30 minutes postoperatively
  Peak expiratory flow (PEF) will be assessed before block and 30 minutes after discharge to Post-Anesthesia Care Unit (PACU) with a laboratory spirometer (Carevusion Germany Spirometer; Master screen PFT). The best value will be measured and recorded
Efficacy of block (Motor) | 30 minutes Postoperatively
  Motor assessment will be tested by using arm abduction (C5), and forearm flexion (C6) (incapacity to overcome gravity= 0; reduced force compared with contralateral arm =1, no loss of force =2). A successful block is defined as motor (score,=0) block in the distribution of the C5 and C6 nerve roots within 30 min of performing the Interscalene Brachial Plexus Block.

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon any reasonable request
Supporting Information: Study Protocol
Time Frame: One year after the end of study